# PROTOCOL TITLE: INTRANASAL INSULIN FOR IMPROVING COGNITIVE FUNCTION IN MULTIPLE SCLEROSIS

DATE: November 20, 2020

**VERSION: 2.4** 

#### **SYNOPSIS**

This will be a randomized, double-blind, placebo-controlled phase I/II pilot study. Participants will be randomized to intranasal insulin 10 international units (IU) twice a day, 20 IU twice a day, or placebo for 24 weeks. Insulin will be administered intranasally using the novel ViaNase<sup>TM</sup> controlled particle dispersion system, allowing for direct delivery of the medication to the nasal epithelium, leading to maximal transport to the CNS (Kurve Technology, Lynnwood, WA).<sup>34</sup> Cognitive assessments will occur at baseline and throughout the 24-week trial, as well as for a period of 24 weeks after discontinuation of the intervention, to evaluate the impact of insulin on cognitive performance as well as the longevity of the treatment response. Biomarkers of cellular stress, neuronal injury, oxidative stress, inflammation, and energy metabolism will be assessed at baseline and at subsequent visits. Stored specimens will be acquired for more detailed future mechanistic studies if intranasal insulin does appear to be safe and effective.

#### INTRODUCTION

Cognitive impairment is common in and devastating to people with MS. MS is a common, chronic, central nervous system (CNS) disease characterized by inflammation, demyelination, and neurodegeneration. One of the most devastating symptoms of this disease is impaired cognitive function, which is common and present in over 60% of individuals with MS. <sup>1-3</sup> MS-related cognitive impairment is associated with lowered quality of life <sup>4</sup> and reduced functional capacity, including loss of employment, <sup>4-7</sup> impaired social relationships, <sup>8</sup> compromised driving safety, <sup>7</sup> and poor adherence to treatment. <sup>9</sup> Impaired cognitive functioning has been observed early in the disease, sometimes even before diagnosis, <sup>10</sup> and cognitive function has been shown to decline longitudinally, both over the short- and long-term. <sup>11-13</sup> Several cognitive domains are impacted in people with MS, including attention, memory, executive functioning, and especially processing speed. <sup>2, 10, 14-18</sup>

To date, multiple pharmacologic interventions have been assessed with disappointing results. There was no significant difference between treatment and placebo for cognition in randomized control trials of donepezil, aminopyridines, gingko biloba, and memantine. Psychostimulants demonstrated some efficacy, but only in secondary outcome measures. Behavioral interventions show promise but are understudied. Furthermore, cognitive rehabilitation is often time consuming, costly, and not universally available. Hence, there is an urgent need to identify or develop novel therapies that can help improve cognitive function in MS.

Insulin is critical for helping with regulation of multiple CNS functions including brain metabolism, neurite outgrowth, neurotransmitter channel activity, neuronal survival, and learning and memory. <sup>25</sup>, <sup>26</sup> There are insulin receptors throughout the brain, with robust concentrations located in eloquent areas including the olfactory bulb, hippocampus, cerebral cortex, and cerebellum. Insulin is present at high levels in the brain and when these levels are decreased, there may be learning and memory impairments. <sup>25</sup>, <sup>27</sup>, <sup>28</sup> The cognitive impairment that can ensue in the context of low brain insulin levels may be related to its ability to protect neurons from various insults including oxidative stress, ischemia, and glutamate-related excitotoxicity. <sup>25</sup>

Moreover, insulin's anti-inflammatory effects, as detailed below, may also impact brain health via suppressing concentrations of chemokines, cytokines, and other molecules that may provoke ongoing CNS inflammation and damage in disease states.

Insulin has biologically relevant anti-inflammatory and neuroprotective CNS effects. At the cellular level, insulin regulates various neuronal functions including receptor expression, trafficking, and survival pathway activation. Insulin signaling in neurons exerts a neuroprotective effect, especially under oxidative stress, via the phosphoinositide-3 kinase (PI3K/AKT) pathway (Figure 1) which, downstream, induces the cAMP response element binding protein (CREB). CREB regulates the expression of several genes that are crucial for learning and memory, including brain derived neurotrophic factor (BDNF),<sup>29</sup> an important promoter of neuronal survival pathways, resulting in regulating learning and memory. This neuroprotective effect has been seen in models of Alzheimer's,



Nature Reviews | Molecular Cell Biology

Parkinson's, and Huntington's Diseases. 30 Insulin also exerts anti-inflammatory effects on peripheral blood

mononuclear cells (PBMCs) by altering inflammatory markers (e.g. monocyte chemoattractant protein-1, chemokine receptor-5) that could ultimately help minimize ongoing nervous system injury.<sup>25</sup>

Insulin's ability to regulate energy metabolism could also result in a protective effect on neurons via impacting oxidative stress and excessive energy demands. Insulin appears to directly mediate brain glucose metabolism maximally within the cortex, and with any disturbance in the communication between insulin and neuronal glucose metabolism, there may be impaired adenosine triphosphate (ATP) synthesis followed by neuronal apoptosis. Moreover, the oxidative stress that results from excessive energy demand leads not only to the production of reactive oxygen species (ROS), but also to ceramide production. These signaling pathways are connected and may be altered upstream by insulin's impact on brain glucose metabolism. For example, several apoptosis-inducing treatments both activate the sphingomyelin (SM)-ceramide pathway and generate oxidative stress. Inflammatory cytokines relevant to MS (e.g. tumor necrosis factor [TNF]- $\alpha$ ) can also induce ceramide formation and ROS. Chemical scavengers prevent elevations in ROS and also SM-ceramide pathway activation. Finally, the use of pyrrolidine dithiocarbamate or N-acetyl cysteine, both antioxidants, restricts ceramide formation and cell death due to TNF- $\alpha$  in rat astrocytes or human breast carcinoma cells.

The impact of insulin in the nervous system, especially as it relates to cognitive health, deserves more attention, as it may be a treatment for disease that cause CNS dysfunction from several pathologies, including MS.

Insulin administration has been shown to improve memory and learning in healthy people and in those with neurodegenerative diseases (see Table 1). Intranasal insulin has shown to have neuroprotective and restorative effects in several human clinical trials. In a recent randomized, double-blind, placebo-controlled study with over 100 people suffering from amnestic mild cognitive impairment or Alzheimer's Disease, intranasal insulin preserved cognitive function in both selective cognitive domains and more globally compared to placebo.<sup>34</sup> The insulin-treated patients also did not show a decline in measures of brain metabolism, whereas the placebo-treated participants did show decreases in fluorodeoxyglucose <sup>18</sup>F uptake in various lobes (parietotemporal, frontal, precuneus, and cuneus). Further, improvements in episodic memory persisted for several weeks after treatment cessation. Overall, these findings suggest that intranasal insulin not only affects cognitive function acutely, but that over time, there may be associated structural changes that lead to a more permanent treatment benefit. Since cognitive dysfunction is very common in MS and can be devastating, a treatment intervention (i.e., intranasal insulin) that can help both acutely and longitudinally is worth pursuing.

Table 1. Summary of past and ongoing human intranasal insulin trials. Adapted from 34-50

| REF. | INTRANASAL<br>INSULIN DOSE | SUBJECTS | ASSESSMENT |
|---|---|---|---|
| Benedict 2004 | 160 IU (long-term) | Healthy | Word list (immediate, delayed recall |
| Reger 2006 | 20 or 40 IU (acute) | Probable AD or MCI vs. healthy | Story recall (immediate, delayed recall) Word list (immediate, delayed recall) |
| Benedict 2007 | 20 IU Aspart vs. 20 IU<br>Regular (long term) | Healthy men | Word list (immediate recall) Word list (delayed recall) |
| Benedict 2008 | 160 IU (acute) | Healthy, normal weight, no meds | Digit span, object location (immediate recall) Mirror tracing (immediate recall) |
| Hallschmid<br>2008 | 160 IU (long-term) | Obese men | Word list (delayed recall) Word list (immediate recall) |
| Reger 2008 | 20 IU (long term) | AD or MCI | Memory score (immediate/ delayed recall ratio) Voice onset time (immediate/delayed recall ratio) |
| Reger 2008 | 10, 20, 40, 60 IU<br>(acute) | AD or MCI<br>vs. healthy | Story recall (immediate recall or delayed recall) Word list learning (immediate & delayed recall) |

| | | | Tippii cation ii. Itaboooyeee i |
|---|---|---|---|
| Krug 2010 | 160 IU (acute) | Healthy women | Digit span (immediate recall) |
| | | | Object location(immediate recall) |
| Fan 2012 | I40 IU (acute) | Schizophrenic | Hopkins Verbal Learning Test |
| <b>Craft 2012</b> | 10 or 20 IU BID | AD or MCI | Verbal Memory Composite |
| Craft 2012 | 20 or 40 IU | AD or MCI | Story recall (delayed recall) |
| McIntyre | 40 IU (long term) | Euthymic with | California Verbal Learning Test, second edition |
| 2012 | | bipolar disorder | Process Dissociation Task |
| <b>Burns 2012</b> | 40 IU (acute) | Early AD | Functional MRI activation; cognitive battery |
| Novak 2013 | 40 IU (long term) | Diabetic | Brief Visuo-spatial Memory Test-Revised |
| | | | Verbal fluency measures |
| Fan 2013 | 40 IU (long term) | Schizophrenic | Cognitive battery |
| Craft 2013 | 20 IU BID | AD or MCI | Cognitive battery |
| <b>Haley 2013</b> | 20 IU | AD | Cerebral glutamate levels; cognitive battery |

AD= Alzheimer's Disease; MCI=mild cognitive impairment; IU=international units; BID=twice daily

Intranasal insulin is extremely safe and tolerable in other populations, allowing for concentrated delivery to the nervous system. Intranasal insulin has a long-standing safety track record that spans more than a decade. *No significant adverse events were reported in the largest intranasal insulin study to date or in any other study that has used intranasal insulin* (see Table 1). An intranasal delivery system provides a non-invasive way to bypass the blood-brain barrier and allow rapid delivery of a medication to the CNS via the olfactory and trigeminal perivascular channels.<sup>34</sup> The main advantage of the delivery system is reducing systemic side effects via limiting a medication's exposure to peripheral organs and tissues. In addition, first-pass metabolism is avoided. Intranasal insulin, as seen in previous human studies, does not adversely affect systemic (blood) glucose or insulin, and it increases CSF insulin to biologically protective concentrations within 30-40 minutes.<sup>51</sup>

# **Intranasal Insulin for Cognition in MS is an Innovative Treatment Approach-Summary**

Insulin appears to activate biologically relevant pathways within the nervous system for regulating and improving learning and memory. The direct and indirect effects of insulin on energy metabolism, oxidative stress, and modulation of inflammatory and neuronal pathways, along with the data from clinical trials in people with other neurodegenerative disorders, prove the rationale for investigating it in people with MS who suffer with cognitive impairment. As noted above, reduced levels of insulin and/or insulin activity may contribute to a number of pathological processes that may ultimately lead to long-term disability in neurodegenerative diseases. Restoring brain insulin to normal levels and increasing insulin sensitivity in the brain may provide therapeutic benefit to people with MS. Herein, we thus propose the first clinical trial in MS to determine the safety and tolerability as well as the effectiveness of intranasal insulin as a therapeutic intervention for cognitive dysfunction. Our study will investigate associated changes in putative biomarkers (see Preliminary Data below) that may corroborate clinical outcomes and provide data regarding the mechanisms by which insulin acts. These measures, along with neuropsychological testing, will be incorporated with safety data in order to accurately assess the potential utility of intranasal insulin for MS cognitive impairment.

#### **OBJECTIVES/AIMS**

Primary Objective: To evaluate the safety and tolerability of intranasal insulin in people with MS

<u>Secondary Objectives:</u> The main secondary objective is to evaluate if intranasal insulin improves cognition in people with MS, as assessed by the SDMT. Additional secondary objectives are to determine if intranasal insulin is associated with changes in additional components of the Minimal Assessment of Cognitive Function in MS (MACFIMS), the Multiple Sclerosis Functional Composite (MSFC) score, health-related quality of life

(Functional Assessment of Multiple Sclerosis [FAMS]), the Expanded Disability Status Scale (EDSS) score, and changes in biomarkers of oxidative stress, neuronal injury, cellular stress, and metabolism.

# Aim 1. To evaluate the safety and tolerability of intranasal insulin in people with MS.

<u>Hypothesis:</u> Intranasal insulin has been shown to be safe in a pilot clinical trial of patients with mild cognitive impairment and Alzheimer's Disease, but its safety and tolerability in MS patients are unknown. We hypothesize that intranasal insulin will be safe and tolerable for people with MS.

# Aim 2. To evaluate if intranasal insulin improves cognition in people with MS.

<u>Hypothesis:</u> Intranasal insulin has been shown to improve multiple aspects of cognition in several randomized, blinded clinical trials of healthy people and in those with mild cognitive impairment and Alzheimer's Disease. We hypothesize that intranasal insulin will improve cognition in MS patients who are cognitively impaired.

# Aim 3. To evaluate the impact of intranasal insulin on measures of oxidative stress, axonal injury, cellular stress, and energy metabolism in MS.

<u>Hypothesis:</u> Although there is not a single biomarker for MS, there are some surrogate measures of interest that may well be impacted by treatment with insulin. We will perform an exploratory analysis to evaluate the effect that intranasal insulin has on these measures, with the hypothesis that *intranasal insulin will improve markers of oxidative and cellular stress, neuronal injury, metabolism, and inflammation in people with MS*.

#### STUDY DESIGN

**Design:** The design of this phase II, randomized, double-blind, placebo-controlled trial is as follows:



**Participants:** The eligibility criteria for the trial are provided in the table below:

| Eligibility Criteria | Rationale |
|---|---|
| Meets 2010 criteria for multiple sclerosis | Study is focused on individuals with MS |
| No relapse in past 3 months | To avoid relapse-induced cognition |
| | confounding |
| Age 18-70 years | To ensure results generalizable |
| At least mild cognitive impairment (1.0 standard deviation | To ensure that we are able to detect |
| or greater below the published mean SDMT z-score, or a | improvements in cognition if insulin does in |
| score of <34 on the processing speed test [PST] | fact have this effect |

| | Application #: IKB00095554 |
|---|---|
| Capacity to learn and self-administer intranasal insulin, or | To ensure that subjects are able to take the |
| presence of a caregiver with such capacity who is willing | medication as prescribed |
| to do it for the duration of the trial | |
| Untreated/on the same MS therapy for at least 2 months, | To avoid change in measures due to change in |
| with no anticipated change in the next year | medication |
| No current, active major depression | May impact results of cognitive testing |
| If on tricyclic antidepressant or anticonvulsant, on stable | May impact results of cognitive testing |
| dose for 6 weeks or more; if on oxybutynin or tolterodine, | |
| on stable dose for > 6 months without plans for changing | |
| dose in next year | |
| If taking selective serotonin (± norepinephrine) reuptake | To minimize impact on cognitive testing |
| inhibitors, pregabalin, gabapentin, sympathomimetic, | without impairing recruitment/limiting |
| monoamine oxidase inhibitor, antipsychotic, amantadine, | generalizability (MS patients use these therapies |
| cholinesterase inhibitor, memantine, modafanil, | commonly) |
| armodafinil, or evening short-acting benzodiazepines, on | |
| stable dose for 6 weeks or greater | |
| Not pregnant or nursing, and willing to prevent pregnancy | Risks of intervention to developing fetus or |
| during study if of childbearing potential | breastfeeding infant unknown |
| No or stable THC use in past 6 weeks; no other illicit drug | To ensure participants can adhere to treatment/ |
| or alcohol abuse in past 3 months* | avoid impact of substances on cognitive testing |
| No known history of diabetes mellitus or insulin resistance | To avoid confounding due to global glucose |
| | dysregulation or use of systemic insulin |
| No active liver disease, stage IV/V kidney disease or | To prevent differential metabolism of insulin |
| severe metabolic derangements | |
| No CNS disorder other than MS or headache | To avoid confounding due to insulin effect on |
| | other disorder |
| No issue making participation not in best interest of patient | To prevent any undue harm to patient |
| During COVID-19 pandemic and related periods of | To ensure minimization of risks to participants |
| slowdown or shutdown, willing to comply with state/local | |
| recommended social distancing and other suggested | |
| COVID-19 related safety measures. Additionally, if female | |
| of childbearing potential, to prevent pregnancy | |

**Recruitment:** Eligible subjects with MS will be recruited from the Johns Hopkins MS Center, at which over 3,000 MS patients, who come from diverse racial/ethnic and socioeconomic backgrounds and from a wide catchment area, are seen annually. We will also screen potentially eligible subjects using an IRB-approved Telephone Screening Script. This will allow us to screen patients who may or may not meet the study's eligibility criteria. If a patient meets the eligibility criteria via telephone screening, we will schedule the patient to come in for a baseline visit. The study coordinator will call only patients of physicians on the study team. Patients interested in participating will be emailed or mailed the written consent form to review in advance.

Since we began routinely administering the iPAD-based correlate of the SDMT, the Processing Speed Test (PST) for all MS Center patients since early 2017 and impaired cognition based on the SDMT is one of the main eligibility criteria, we will quickly be able to focus recruitment efforts on those who have evidence of mild cognitive impairment, eliminating the need for an extra screening visit. More than 80 people with MS who are currently enrolled in various studies in the center already have SDMT data and thus will also be easily screened

for eligibility, even if they haven't had a recent clinic visit. For MS Center patients that have not taken an SDMT or PST test, we will use an oral consent process to administer the SDMT test and determine eligibility. SDMT or PST test results obtained within 3 months of the baseline visit will be considered as proof of eligibility for the study and may be screened in person or by phone. The study coordinator will only approach MS Center patients of physicians on the study team or those referred by their treating physician. In addition to the above recruitment strategies, we will obtain home-based PST screening test for our MS patients that have iPADs (Air, Air 2, and iPAD 2017), as the PST app is now available. This will allow for remotely screening potential subjects that have transportation and/or mobility limitations. If at any time point, enrollment is less than 85% of the target, we will interview subjects who have declined to participate to determine the deterrents to enrollment; we will then implement alterations in recruitment needed to enhance enrollment.

Study Treatment: Intranasal insulin (Novolin R, Novo Nordisk, Princeton, NJ) will be evaluated in two doses (10 IU twice a day, 20 IU twice a day) and compared to the sterile diluent (Eli Lilly and Company – NDC:00002-0800) (1:1:1 randomization, stratified by relapsing versus progressive MS). The 20 IU dose will consist of insulin. The 10 IU dose will be a diluted mixture comprised of normal saline and insulin. The study drug, insulin, has a distinct smell. In order to preserve study blinding, we will use the Lilly sterile diluent, which has a similar odor as the insulin, to preserve blinding. The study drug and placebo (Lilly diluent) will be prepared by the Johns Hopkins Investigational Drug Service and will appear identical to maintain blinding. A nasal drug delivery device (Kurve Technology, Lynnwood, WA) will be utilized to ensure optimal exposure of the olfactory epithelium. The treatment regimen was chosen to match that of a recent successful pilot study in Alzheimer's Disease. <sup>34</sup> Evaluating two doses will allow for the possibility that any benefit of insulin may be non-linear.

<u>Treatment Preparation</u>: The study pharmacist will transfer either insulin; sterile diluent (placebo); or normal saline into 10cc empty syringes to preserve study blinding. The syringes will be labeled syringe A or syringe B, respectively. At the baseline visit, subjects and/or caregivers will be instructed on how to fill the cartridges by adding one A and one B syringe to the cartridge; gently mix the contents and be shown how to administer the doses using the ViaNase device. Due to the 28-day shelf life of the insulin/diluent, the subjects need to know how to refill their own study products prior to their next study visit.

Methods to Maximize Adherence: Given data from prior studies, it is anticipated that adverse events will not reduce adherence. The study coordinator will help each participant set reminder alarms on watches or phones; those who do not have access to such devices will be given a medication alarm watch for use during the study. Study staff will also identify a patient advocate and to educate that person to help the study participant maintain adherence. To maximize visit adherence, patients will receive a reminder in the week prior to the appointment.

Accountability of Medication: A sufficient amount of medication will be supplied at the baselineand week 12 visits to ensure the supply will last until the next study visit, otherwise, refills will be mailed to the participants. Participants will be asked to return unused medication at each study visit for adherence assessment. The Johns Hopkins Investigational Drug Unit will maintain adequate records of the disposition of the study drug and accounts of any destroyed study drug.

**Study Personnel:** All personnel (except the statistician) will be blinded to treatment assignment. The <u>treating physician</u> will assess eligibility criteria, obtain informed consent, obtain and maintain the medical history and medication record, monitor patients' safety, conduct the physical examination, and evaluate and report adverse events. The <u>examining physician</u> will perform the blinded EDSS. The blinded <u>study neuropsychologist</u> will administer the MACFIMS to participants. The blinded <u>study coordinator</u> will be responsible for the study's administrative duties, obtaining vital signs, conducting the MSFC and administering the depression, suicidality, and health-related quality of life measures, and drawing and processing blood samples as well as urine

pregnancy testing, when indicated. The <u>laboratory technician</u> will conduct the biomarker analyses for Aim 3. <u>Other personnel</u> include Drs. Haughey and Calabresi, who will interpret biomarker data. A statistician from the Johns Hopkins School of Public Health will create the randomization schedule and perform final data analyses.

**Study Visits:** The visit schedule is detailed below. Visits will take place within  $\pm 5$  days of the target date.

| | Week 0 | Week 6 | Week 12 | Week 24 | Week 36 | Week 48 |
|---|---|---|---|---|---|---|
| Written consent | X | | | | | |
| Verify eligibility | X | | | | | |
| Teaching and First dose | X | | | | | |
| administration and observation | | | | | | |
| Medical history, relapse assessment | X | X | X | X | X | X |
| Medication review | X | X | X | X | X | X |
| Vital signs | X | X | X | X | X | X |
| Physical, neurologic (EDSS) exams | X | | X* | X* | | X* |
| MS Functional Composite | X | X | X | X | X | X |
| Adverse event assessment | | X | X | X | X | X |
| Biomarker evaluation | X | X | X | X | X | X |
| Stored blood for future studies | X | X | X | X | X | X |
| DXA scan | X | | | | | |
| A pregnancy test (if woman of | X | X | X | X | | |
| childbearing potential) | | | | | | |
| MACFIMS battery | X | | X | X | X | X |
| Sleep questionnaires | X | | X | X | | X |
| Depression and quality of life | X | X | X | X | X | X |
| Suicidality evaluation | X | X | X | X | X | X |

<sup>\*</sup>EDSS only

Schedule Modification during COVID-19 (will be in effect unless JHU operations have returned to normal, a COVID-19 vaccine has been developed, or evidence of substantial likelihood of herd immunity from COVID-19 due to a high proportion of previously-infected individuals). Additionally, due to COVID-19 and staffing shortages during the holiday season, we will allow study visits within  $\pm$  10 days of the target date if needed to ensure the safety of the participants.

| | Week 0 | Week | Week | Week 24 | Week | Week 48: |
|---|---|---|---|---|---|---|
| | | 6: | 12** | | 36: | Virtual% |
| | | Virtual | | | Virtual | |
| Written consent& | X | | | | | |
| Verify eligibility | X | | | | | |
| Teaching and First dose | X | | | | | |
| administration and observation | | | | | | |
| Medical history, relapse | X | X | X | X | X | X |
| assessment | | | | | | |
| Medication review | X | X | X | X | X | X |
| Vital signs | X | | X | X | | |
| Neurologic (EDSS) exam | X | | | | | |
| MS Functional Composite | X | | X*** | X*** | | |

| Adverse event assessment | | X | X | X | X | X |
|---------------------------------|-----|---|-----|-----|---|---|
| Biomarker evaluation | X | | X | X | | |
| Stored blood for future studies | X\$ | | X\$ | X\$ | | |
| DXA scan | X | | | | | |
| Pregnancy assessment* | X* | X | X | X | | |
| MACFIMS battery | X | | X | X | | X |
| Sleep questionnaires | X | | X | X | | X |
| Depression and quality of life | X | X | X | X | X | X |
| Suicidality evaluation | X | X | X | X | X | X |

<sup>\*</sup>Pregnancy test at baseline; document last menstrual period/adequate pregnancy prevention plan at virtual follow-ups (for women of childbearing potential)

% if COVID-19 pandemic is lifted, we will still complete this visit in-person; we will accept a study window that extends 3 months beyond week 48 if there is indication at that time, even if the pandemic is still affecting safety, that it will soon be safe again (e.g. vaccine developed or clear evidence of critical percentage of population has already been infected, fully operational at JHU)

If a severe COVID-19 outbreak occurs again such as occurred in the spring of 2020, we will conduct all follow-up assessments by video or phone until such time as it is safe to pursue the modified schedule, as above, or resume the originally-planned schedule.

All study visits will be scheduled for the morning to reduce variability in cognitive function related to the time of day. At baseline, fasting laboratory testing will be performed, including a hemoglobin A1c test and insulin level. All subjects will then be given breakfast prior to completing cognitive testing. For follow-up visits, all subjects will complete the MACFIMS battery after eating a usual meal (if the participant came without having eaten, breakfast will be provided to them) and prior to taking the morning dose of study treatment. Unscheduled visits will occur if any safety issue arises.

In order to ensure subjects (or their responsible caregivers) are able to use the medication as instructed, all subjects and caregivers (when relevant) will be instructed on the use of the inhaler and will be observed by a health care provider when performing their first dose administration at the time of the first visit.

#### Risks

#### Intranasal insulin

Intranasal insulin has been shown to be safe and tolerable in other populations and patient groups, but it has never been studied in people with MS. The most common side effects related to irritation of the nasal passages. Giving insulin through the nose did not result in lower circulating glucose levels in other studies, but the first 15

<sup>\*\*</sup>will convert to virtual follow-up with activities equal to week 6 if stay-at-home orders recur Items that are in **bold** will be done either virtually or in-person until operations are fully normalized with respect to COVID-19 pandemic; in addition, some aspects of the MACFIMS neuropsychological battery can (and will) be done virtually as well

<sup>\*\*\*</sup>timed 25-foot walk only

<sup>&</sup>amp;Consent will be reviewed at length virtually within the week prior to the day of the visit, with all questions asked at that time. At the baseline visit, patients will be given the opportunity to ask any remaining questions and can sign during the teleconsent, if capable, or will sign at the time of the baseline visit.

people in this study will be monitored for this potential risk by testing a fingerstick blood glucose level periodically for 90 minutes after the first dose of intranasal insulin (see <u>Safety</u> section under **Outcomes** on page 10).

Insulin, given by the more traditional subcutaneous route, has the following potential risks:

Hypoglycemia: Common symptoms of hypoglycemia include sweating, dizziness or lightheadedness, shakiness, hunger, a fast heartbeat, tingling of the hands, feet, lips or tongue, trouble concentrating, confusion, blurry vision, slurred speech, anxiety, irritability, or mood changes, or headache. Very low blood sugar can cause loss of consciousness, seizures, or temporary or permanent brain problems or death. Mild hypoglycemia can be treated by drinking or eating something sugary right away (fruit juice, sugar candies, or glucose tablets).

Hypokalemia: Hypokalemia can lead to breathing problems, low heartbeat, or death.

Allergic reaction: Common symptoms of an allergic reaction include a rash all over the body, trouble breathing, a fast heartbeat, sweating, and feeling faint.

Weight gain or swelling of the arms and legs.

While these are all risks potentially associated with subcutaneous administration of insulin, none of these risks has been demonstrated to be the case in the published trials of intranasal insulin. Thus, by avoiding the traditional route of administration, it is anticipated that these risks will be minimized.

#### **Blood Draw**

Taking blood may cause discomfort, bleeding or bruising where the needle enters the body. In rare cases, it may result in fainting. There is a small risk of infection. To minimize the risks, blood will be drawn by a trained study team member/phlebotomist.

#### Confidentiality

Despite the best efforts of the research team, there may still be a risk if information about participants were to become known to people outside of this study.

# **Questionnaires**

Participants may get tired or bored when we are asking questions or they are completing questionnaires. They do not have to answer any question they do not want to answer.

# **DXA** scan

DXA testing is painless and involves exposure to radiation. This research study includes exposure to radiation from x-rays or gamma rays. This radiation exposure is for research purposes only and is not part of the participant's medical care. X-rays and gamma rays can damage cells, but at low doses, the body is usually able to repair these cells.

The radiation exposure that participants will get in this research study is 0.001 rem. This is less than the 0.3 rem that the average person in the United States gets each year from natural sources like the sun, outer space, air, food, and soil. The risk from the radiation exposure in this research study is very small. The radiation exposure described here is what participants will get from this research study only. It does not include any exposure

participants may have received or will receive from other medical tests outside of this study that are a part of their medical care.

### **Benefits**

There is no known benefit of intranasal insulin, and thus there is no known risk of being in the placebo group. All patients who are already on a medication for MS will be allowed to continue that medication during the study.

# **Payment and Remuneration**

Participants will receive a parking coupon at each visit.

### **Costs**

There are no costs to participants for taking part in this study.

#### **Outcomes:**

<u>Safety</u> Since this medication was extremely well-tolerated in several published studies, <sup>34-50</sup> we anticipate the same will be true for people with MS. In prior studies, there was no effect of intranasal insulin on serum glucose levels. However, we will monitor the first 15 participants for a period of 90 minutes after their first dose of the medication to evaluate serial finger stick blood glucose levels. If there is a clinically significant reduction in these levels, we will convene a Data Safety Monitoring Board (DSMB) meeting to adjust the protocol. We will also record and, when appropriate, report all patient-reported adverse events, as described below. Subjects and their caregivers will be required to keep an electronic diary of adverse events, which will be reviewed at each study visit. As mandated by the FDA, the Columbia Suicide Severity Rating Scale will be administered at each study visit.

Cognitive Assessments The MACFIMS battery includes the following: The Symbol Digit Modalities Test (SDMT) is commonly used in MS to assess processing speed.<sup>1, 52-54</sup> The oral version of the test is recommended for MS since the written version may be confounded by upper extremity weakness.<sup>53, 55, 56</sup> There are three alternate versions of this test with strong psychometric properties.<sup>37</sup> A 3.5-4 point raw score difference on the SDMT has been identified as clinically meaningful.<sup>6, 57</sup> The Controlled Oral Word Association Test (COWAT) measures phonemic fluency.<sup>58</sup> The California Verbal Learning Test, Second Edition (CVLT-II) is a verbal learning and memory test.<sup>55, 59</sup> The Brief Visuospatial Memory Test – Revised (BVMT-R) is a visual, nonverbal test of learning and memory.<sup>60</sup> The Rao-version of the Paced Auditory Serial Addition Test (PASAT) evaluates processing speed, working memory, and basic addition skills.<sup>58</sup> Visual-spatial abilities are assessed with the Judgement of Line Orientation Test (JLO).<sup>58, 61</sup> The Delis-Kaplan Executive Function System (DKEFS) tests executive functioning, concept formation, and cognitive flexibility.

**Exploratory Biomarkers** Plasma and/or PBMCs will be collected at baseline, week 12, and week 24 visits (except if COVID-19 related shutdown does not permit follow-up blood collection or lab-based processing) and will be isolated and cryopreserved for batch analyses in the labs of Dr. Haughey or Calabresi. Inflammatory (cytokines, lymphocyte subsets), metabolic (Kreb's cycle substrate, fatty acids), cellular stress (ceramides, sphingomyelin) and neurotrophic (BDNF) measures, as well as markers of oxidative stress (protein carbonyls, 8-isoprostane, nitrotyrosine, and 4-hydroxynonenal adducts [lysine and histidine]), will be quantified. Since our data show oxidative stress biomarkers and elevated ceramides in plasma of MS patients and recent work shows

the brain has lymphatics, explaining how brain metabolites return to the periphery, blood biomarkers are a relevant and convenient way to monitor CNS metabolism.<sup>62</sup>

Additional Outcomes and Assessment of Covariates In order to identify and, if needed, adjust for comorbid depression, the Beck Depression Inventory will be administered at each study visit. Health-related quality of life will also be assessed utilizing the FAMS. We will also evaluate how overall sleep quality in people with MS impacts health-related quality of life. We will also evaluate for occult insulin resistance or differences in metabolism in several ways. We will evaluate dual-energy x-ray absorptiometry (DXA) at baseline, which will help determine body composition, in particular bone density. We will also calculate an insulin resistance index, the homeostatic model assessment (HOMA-IR),<sup>63</sup> using baseline fasting glucose and insulin. Statistical models exploring these body composition and insulin resistance parameters as potential confounders or mediators will be evaluated. Finally, the MACFIMS, safety, depression, and health-related quality of life outcomes will be monitored after discontinuation of the insulin (or placebo) to evaluate for any decline in cognitive function associated with medication discontinuation.

Safety/Adverse Event Monitoring An adverse event (AE) is any occurrence or worsening of an undesirable or unintended sign, symptom (or abnormal laboratory test), or disease temporally associated with the use of a medicinal product or intervention, whether or not it is considered related to the product/intervention. We will use the National Cancer Institute's Common Terminology Criteria for Adverse Events version 4.0 to report and grade all adverse events, whether or not they are related to disease progression or treatment. The relationship between an AE and the intervention will be determined by the blinded study physician and recorded on the appropriate form. The investigator will record all study adverse events in the chart and will treat participants with AEs appropriately, observing them until they resolve or stabilize. AEs will be collected from the start of the study until a participant terminates from the study; those that are unresolved at the time of termination will be followed until they resolve or up to 30 days. An adverse event is considered unexpected when its nature or severity is not consistent with the product information (e.g. protocol or the informed consent form). Serious AEs will be collected from informed consent signing until 30 days after study completion or until 30 days after a participant withdraws from the study. The following process for reporting a serious AE will ensure compliance with the International Conference on Harmonisation guidelines: the Institutional Review Board (IRB) and DSMB will be notified in two business days of a serious AE that is medication-related and unexpected, and standard reporting (15 calendar days) will occur if the event is serious, expected and medication-related, serious, expected and not medication-related, or serious, unexpected and not medicationrelated. Life-threatening events will be reported within 7 calendar days. Any pregnancy will be reported to the IRB and DSMB, and pregnancies will be followed to their conclusion. Female participants who become pregnant will stop the study intervention. The investigator will report pregnancies to the IRB within two business days. The study medication will be discontinued if an AE grade 3 or higher occurs and is at least possibly related to the medication or if the subject cannot tolerate the medication/ wants to discontinue it. Any death that is at least possibly related to the study will put the study on hold until the DSMB evaluates it.

<u>DSMB</u>: The DSMB consists of an independent neurologist, an endocrinologist, and a statistician. It will convene any time an adverse event ≥ grade 3 occurs and routinely at 25%, 50%, 75%, and 100% enrollment. All serious adverse events will be promptly and simultaneously reported to the IRB, the DSMB and the Independent Research Monitor. Only serious adverse events (SAEs) that would also meet the definition of an Unanticipated Problem Involving Risks to Subjects or Others (UPIRTSOs) that are related to the protocol will be promptly reported to the United States Army Medical Research and Materiel Command Office of Research Protections Human Research Protection Office HRPO (USAMRC ORP HRPO).

<u>Independent Research Monitor:</u> The PI, Dr. Mowry, has appointed Dr. Anne Damian, a trained neurologist, as the Independent Research Monitor. Dr. Damian will provide independent safety review and will have the

authority to stop the research study; remove an individual subject from the research study; and will take any steps to protect the safety and well-being of the subjects until the IRB can assess the problem or event. The independent research monitor must review all unanticipated problems involving risks to subjects or others (UPIRTSO), but not all SAEs. The monitor will review the SAEs if they also meet the definition of a UPIRTSO and will provide an unbiased written report of the event. The Research Monitor will comment on the outcomes of the event or problem and the relationship to participation in the study. Additionally, the research monitor will indicate whether she concurs with the details of the report provided by the principal investigator.

# **Analytic Plan**

**Aim 1.** Safety data will be analyzed as they are captured in real time. Assessments will focus on AEs (including study treatment tolerability assessments, laboratory evaluations, vital signs, and physical examination). The incidence rate of AEs will be recorded by system organ class, severity, and by relationship to the study treatment. Tolerability analysis will be based on the number (%) of subjects who failed to complete the study due to adverse events. Lab values for each parameter will be summarized by shift tables. For quantitative parameters, summary statistics for actual values and change from baseline will be presented. Changes in the first 24 weeks will be compared between groups using mixed effects regression analyses to account for the longitudinal nature of the data using random subject-specific intercepts and slopes.

Aim 2. Summary statistics (mean ± standard deviation, median and interquartile range, or number and percentages) will be used to characterize the outcomes. For each cognitive outcome, to evaluate variability in the estimated means across groups, assuming that the within-group means are normally distributed, a one-way ANOVA will be conducted at the follow-up visits during the first 24 weeks. If the within-group data are strongly non-Gaussian, a Kruskal-Wallis test will be used. A mixed effects longitudinal model will also be used to test whether any differences across groups exist at the follow-up visits within the first 24 weeks. Further, models accounting for covariates of interest, including the HOMA-IR, body composition, body mass index, age, sex and depression, will be evaluated. For within-person changes in measures at follow-up compared to baseline, paired t-tests will be used. We will also evaluate the SDMT at each study visit and other MACFIMS outcomes at week48 to establish the longevity of any therapeutic response to insulin.

**Aim 3.** For the biomarker outcomes, to evaluate variability in the estimated means across groups, assuming that the within-group means are normally distributed, a one-way ANOVA will be conducted at the follow-up visits during the active treatment phase. If the within-group data are strongly non-Gaussian, a Kruskal-Wallis test will be used. A mixed effects longitudinal model will also be used to test if differences across groups exist at follow-up visits. For within-person changes in measures at follow-up compared to baseline or before versus after calorie restriction days, paired t-tests will be used. Correlations between the biomarkers will be assessed. A bootstrap of subjects will be used to obtain 95% equal confidence intervals for these measures. We will also evaluate the biomarker changes after study therapy ends.

**Sample Size and Power:** Sample size estimates are difficult given the novelty of the project but are based on the goal of detecting a benefit of insulin on cognition. In a pivotal study of two doses of intranasal insulin versus placebo in participants with mild cognitive impairment or mild to moderate Alzheimer's Disease, the Dementia Severity Rating Scale score improved over the four-month treatment course in those receiving intranasal insulin.<sup>34</sup> Using the scores in the 10 IU twice a day group, given a two-sided alpha of 0.05 and beta 0.20 (80% power), assuming 3 follow-up cognitive tests and a correlation between baseline and follow-up results of 0.5, 29 subjects per group are required. To account for drop-outs and for the three-arm design, a total of 35 subjects per group is planned. With SDMT as the outcome, for a two-arm design, this sample size confers 80% power (assuming SDMT standard deviation of 9 points and two-sided alpha of 0.05) to detect a 6-point improvement in SDMT which seems reasonable considering that transcranial stimulation with cognitive training

improved SDMT by an average of more than 8 points compared to cognitive training alone in a pilot study of 20 subjects. We do not expect that this study will provide conclusive evidence of efficacy for cognition, but it will provide estimates of the mean and standard deviation of the distribution in change in cognitive tests that will inform the design of definitive, phase III trials. Aim 3 is exploratory, but given the relative abundance differences in MS versus controls in our preliminary data in C22:1, and assuming a similar absolute C22:1 concentration as in women aged 55-64 years, with 35 subjects in a two-arm study of 35 subjects/arm and a 2-sided alpha of 0.05, we will have 80% power to detect a 10 ng/mL difference in ceramide levels.

#### REFERENCES CITED

- 1. Benedict RH, et al. Validity of the minimal assessment of cognitive function in multiple sclerosis (MACFIMS). J Int Neuropsychol Soc 2006;12:549-558.
- 2. DeLuca J. What we know about cognitive changes in multiple sclerosis. In: LaRocca N, Kalb R, eds. Multiple Sclerosis: Understanding the Cognitive Challenges. New York: Demos Health; 2006: 17-40.
- 3. Rao S. Cognitive Function in Patients with Multiple Sclerosis: Impairment and Treatment. IJMSC 2004;1:9-22.
- 4. Ruet A, Deloire M, Hamel D, Ouallet JC, Petry K, Brochet B. Cognitive impairment, health-related quality of life and vocational status at early stages of multiple sclerosis: a 7-year longitudinal study. J Neurol 2013;260(3):776-84.
- 5. Strober LB, Christodoulou C, Benedict RH, Westervelt HJ, Melville P, Scherl WF et al. Unemployment in multiple sclerosis: the contribution of personality and disease. Mult Scler 2012;18(5):647-53.
- 6. Morrow SA, Drake A, Zivadinov R, Munschauer F, Weinstock-Guttman B, Benedict RH. Predicting loss of employment over three years in multiple sclerosis: clinically meaningful cognitive decline. Clin Neuropsychol 2010;24(7):1131-45.
- 7. Schultheis MT, Weisser V, Ang J, Elovic E, Nead R, Sestito N et al. Examining the relationship between cognition and driving performance in multiple sclerosis. Arch Phys Med Rehabil 2010;91(3):465-73.
- 8. Patti F. Optimizing the benefit of multiple sclerosis therapy: the importance of treatment adherence. Patient Prefer Adherence 2010;4:1-9.
- 9. Chiaravalloti ND, DeLuca J. Cognitive impairment in multiple sclerosis. Lancet Neurol 2008; 7(12):1139-1151.
- 10. Rao SM et al. Cognitive dysfunction in multiple sclerosis. II. Impact on employment and social functioning. Neurology. 1991;42:692-696.
- 11. Amato MP, Razzolini L, Goretti B, Stromillo ML, Rossi F, Giorgio A et al. Cognitive reserve and cortical atrophy in multiple sclerosis: a longitudinal study. Neurology 2013;80(19):1728-33.
- 12. Amato MP, Ponziani G, Siracusa G, Sorbi S. Cognitive dysfunction in early-onset multiple sclerosis: a reappraisal after 10 years. Arch Neurol 2001;58(10):1602-6.
- 13. Lacy M, Hauser M, Pliskin N, Assuras S, Valentine MO, Reder A. The effects of long-term interferon-beta-1b treatment on cognitive functioning in multiple sclerosis: a 16-year longitudinal study. Mult Scler 2013;19(13):1765-72.
- 14. Deluca J, Barbieriberger S, Johnson SK. The nature of memory impairments in multiple sclerosis-acquisition versus retrieval. Journal of Clinical and Experimental Neuropsychology 1994;16(2):183-9.
- 15. DeLuca J, Gaudino EA, Diamond BJ, Christodoulou C, Engel RA. Acquisition and storage deficits in multiple sclerosis. Journal of Clinical and Experimental Neuropsychology 1998;20(3):376-90.
- 16. Thornton AE, Raz N, Tucker KA. Memory in multiple sclerosis: Contextual encoding deficits. Journal of the International Neuropsychological Society 2002;8(3):395-409.

- 17. DeLuca J, Chelune GJ, Tulsky DS, Lengenfelder J, Chiaravalloti ND. Is speed of processing or working memory the primary information processing deficit in multiple sclerosis? J Clin Exp Neuropsychol 2004;26(4):550-62.
- 18. Demaree HA, DeLuca J, Gaudino EA, Diamond BJ. Speed of information processing as a key deficit in multiple sclerosis: implications for rehabilitation. J Neurol Neurosurg Psychiatry 1999;67(5):661-3.
- 19. Krupp LB, et al. Multicenter randomized clinical trial of donepezil for memory impairment in multiple sclerosis. Neurology. 2011;76(17):1500-1507.
- 20. Solari A, Uitdehaag B, Giuliani G, Pucci E, Taus C. Aminopyridines for symptomatic treatment in multiple sclerosis. Cochrane Database Syst Rev 2001(4):Cd001330.
- 21. Lovera JF, Kim E, Heriza E, Fitzpatrick M, Hunziker J, Turner AP et al. Ginkgo biloba does not improve cognitive function in MS: a randomized placebo-controlled trial. Neurology 2012;79(12):1278-84.
- 22. Lovera JF, Frohman E, Brown TR, Bandari D, Nguyen L, Yadav V et al. Memantine for cognitive impairment in multiple sclerosis: a randomized placebo-controlled trial. Mult Scler 2010;16(6):715-23.
- 23. Morrow SA, Kaushik T, Zarevics P, Erlanger D, Bear MF, Munschauer FE et al. The effects of L-amphetamine sulfate on cognition in MS patients: results of a randomized controlled trial. J Neurol 2009;256(7):1095-102.
- 24. Mitolo M, Venneri A, Wilkinson ID, Sharrack B. Cognitive rehabilitation in multiple sclerosis: A systematic review. J Neurol Sci 2015;354(1-2):1-9.
- 25. Duarte AI, Moreira PI, Oliveira CR. Insulin in Central Nervous System: More than Just a Peripheral Hormome. J Aging Res. 2012;2012:384017.
- 26. Apostolatos A, Song S, Acosta S, et al. Insulin promotes neuronal survival via the alternatively spliced protein kinase CδII isoform. J Biol Chem 2012 Mar 16;287(12):9299-310.
- 27. Schechter R, Whitmire J, Holtzclaw L, George M, Harlow R, Devaskar SU. Developmental regulation of insulin in the mammalian central nervous system. *Brain Research*, vol. 582, no. 1, pp. 27–37, 1992.
- 28. LeRoith E. CNS regulation of carbohydrate metabolism in *Advances in Metabolic Disorders*, A. Szabo, Ed., vol. 10, pp. 304–340, Academic Press, 1983.
- 29. Altarejos JY, Montminy M. CREB and the CRTC co-activators: Sensors for hormonal and metabolic signals. Nat Rev Mol Cell Biol 2011;12:141-151.
- 30. Duan W, Guo Z, Jiang H, Ware M, Li XJ, Mattson MP. Dietary restriction normalizes glucose metabolism and BDNF levels, slows disease progression, and increases survival in huntingtin mutant mice. Proc Natl Acad Sci U S A 2003;100:2911-2916.
- 31. Bingham EM, Hopkins D, Smith D et al. The role of insulin in human brain glucose metabolism: an 18fluorodeoxyglucose positron emission tomography study. Diabetes 2002;51:3384-3390.
- 32. Russell JW, Golovoy D, Vincent AM, et al. High glucoseinduced oxidative stress and mitochondrial dysfunction in neurons. FASEB J 2002;16:1738–1748.
- 33. Andrieu-Abadie N, Gouaze V, Salvayre R, Levade T. Ceramide in apoptosis signaling: relationship with oxidative stress. Free radical biology & medicine 2001;31:717-728.
- 34. Craft S, Baker LD, Montine TJ, et al. Intranasal insulin therapy for Alzheimer Disease and amnestic mild cognitive impairment. Arch Neurol 2012;69:29-38.
- 35. Benedict C, Hallschmid M, Hatke A, et al. Intranasal insulin improves memory in humans. Psychoneuroendocrinology 2004;29:1326-1334.
- 36. Benedict C, Hallscmid M, Schmitz K, et al. Intranasal insulin improves memory in humans: superiority of insulin aspart. Neuropsychopharmacology 2007;32:239-243.
- 37. Benedict C, Kern W, Schultes B, Born J, Hallschmid M. Differential sensitivity of men and women to anorexigenic and memory-improving effects of intranasal insulin. J Clin Endocrinol Metab 2008;93:1339-1344.

- 38. Hallschmid M, Benedict C, Schultes B, Born J, Kern W. Obese men respond to cognitive but not to catabolic brain insulin signaling. Int J Obes 2008;32:275-282.
- 39. Reger MA, Watson GS, Frey WH, et al. Effects of intranasal insulin on cognition in memory-impaired older adults: modulation by APOE genotype. Neurobiol Aging 2006;27:451-458.
- 40. Reger MA, Watson GS, Green PS, et al. Intranasal insulin improves cognition and modulates beta-amyloid in early AD. Neurology 2008;70:440-448.
- 41. Reger MA, Watson GS, Green PS, et al. Intranasal insulin administration dose-dependently modulates verbal memory and plasma amyloid-beta in memory-impaired older adults. J Alzheimers Dis 2008;13:323-331.
- 42. Krug R, Benedict C, Born J, Hallschmid M. Comparable sensitivity of postmenopausal and young women to the effects of intranasal insulin on food intake and working memory. J Clin Endocrinol Metab 2010;95:E468-E472.
- 43. Fan X, Copeland PM, Liu EY, et al. No effect of single-dose intranasal insulin treatment on verbal memory and sustained attention in patients with schizophrenia. J Clin Psychopharmacol 2011;31:231-234.
- 44. Fan X, Liu E, Freudenreich O, et al. No effect of adjunctive, repeated-dose intranasal insulin treatment on psychopathology and cognition in patients with schizophrenia. J Clin Psychopharmacol 2013;33:226-230.
- 45. McIntyre RS, Soczynska JK, Woldeyohannes HO, Miranda A, Vaccarino A, Macqueen G, Lewis GF, Kennedy SH. A randomized, double-blind, controlled trial evaluating the effect of intranasal insulin on neurocognitive function in euthymic patients with bipolar disorder. Bipolar Disord 2012;14:697-706.
- 46. https://www.clinicaltrials.gov/ct2/show/NCT01547169?term=intranasal+insulin+verbal+memory&rank=1. Accessed July 30, 2015.
- 47. https://www.clinicaltrials.gov/ct2/show/NCT00581867?term=intranasal+insulin+burns&rank=1. Accessed July 30, 2015.
- 48. Novak V, Milberg W, Hao Y, et al. Enhancement of vasoreactivity and cognition by intranasal insulin in type 2 diabetes. Diabetes Care 2014;37:751-759.
- 49. https://www.clinicaltrials.gov/ct2/show/NCT01595646?term=craft+intranasal+insulin&rank=3. Accessed July 30, 2015.
- 50. https://www.clinicaltrials.gov/ct2/show/NCT01145482?term=intranasal+insulin+haley&rank=1. Accessed July 30, 2015.
- 51. Born J, Lange T, Kern W, McGregor GP, Bickel U, Fehm HL. Sniffing neuropeptides: A transnasal approach to the human brain. Nat Neurosci 2002;5:514-516.
- 52. D'hooghe MB, Cleynhens K, D'hooge M, Haelewyck MC, DeKeyser J, Nagels G. The Symbol Digit Modalities Test as a sentinel test for cognitive impairment. Eur J Neurol 2014;21:1219-1225.
- 53. Benedict RH, Duquin JA, Jurgensen S, Rudick RA, Feitcher J, Munschauer FE et al. Repeated assessment of neuropsychological deficits in multiple sclerosis using the Symbol Digit Modalities Test and the MS Neuropsychological Screening Questionnaire. Mult Scler 2008;14(7):940-6.
- 54. Benedict RH SA, Parikh R, Rodgers J, Cadavid D, Erlanger D. Reliability and equivalence of alternate forms for the Symbol Digit Modalities Test: implications for multiple sclerosis clinical trials. Mult Scler 2012;18(9):1320-5.
- 55. Langdon DW, Amato MP, Boringa J, Brochet B, Foley F, Fredrikson S et al. Recommendations for a Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS). Mult Scler 2012;18(6):891-8.
- 56. Brochet B, Deloire MS, Bonnet M, Salort-Campana E, Ouallet JC, Petry KG et al. Should SDMT substitute for PASAT in MSFC? A 5-year longitudinal study. Mult Scler 2008;14(9):1242-9.
- 57. Benedict RH, Morrow S, Rodgers J, Hojnacki D, Bucello MA, Zivadinov R et al. Characterizing cognitive function during relapse in multiple sclerosis. Mult Scler 2014;20(13):1745-52.
- 58. Benedict RH FJ, Archibald CJ, Arnett PA, Beatty WW, Bobholz J, Chelune GJ, Fisk JD, Langdon DW, Caruso L, Foley F, LaRocca NG, Vowels L, Weinstein A, DeLuca J, Rao SM, Munschauer F. Minimal

- neuropsychological assessment of MS patients: a consensus approach. Clin Neuropsychol 2002;16(3):381-97.
- 59. Panou T, Mastorodemos V, Papadaki E, Simos PG, Plaitakis A. Early signs of memory impairment among multiple sclerosis patients with clinically isolated syndrome. Behav Neurol. 2012;25(4):311-26.
- 60. Benedict R. Brief Visuospatial Memory Test-Revised: Professional manual. Lutz, FL: Psychological Assessment Resources, Inc.
- 61. Benton AL, Sivan AB, Hamsher Kd, Varney NR, Spreen O. Contributions to Neuropsychological Assessment: A Clinical Manual. Oxford University Press; 1994.
- 62. Louveau A, Smirnov I, Keyes TJ et al. Structural and functional features of central nervous system lymphatic vessels. Nature 2015;523:337-341.
- 63. Willette AA, Bendlin BB, Starks EJ, et al. Association of insulin resistance with cerebral glucose uptake in late middle-aged adults at risk for Alzheimer Disease. JAMA Neurol 2015 (in press).
- 64. Mattioli F, Bellomi F, Stampatori C, Capra R, Miniussi C. Neuroenhancement through cognitive training and anodal tDCS in multiple sclerosis. Mult Scler J 2015 (in press).
- 65. Mielke MM, bandaru VV, Han D, et al. Demographic and clinical variables affecting mid- to late-life trajectories of plasma ceramide and dihydroceramide species. Aging Cell 2015 (in press).

# **Trial Protocol for:**

Intranasal Insulin for Improving Cognitive Function in Multiple Sclerosis (NCT02988401)

Date of Protocol 11/20/2020